CLINICAL TRIAL: NCT02042716
Title: Added Value of Supersonic Shear Imaging in the Diagnosis of White Matter Damage in Preterm Infants
Acronym: BELUGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P120601; ID RCB : 2012-A01530-43 (Other: ID RCB)
Record Dates: First submitted 2013-07-26; First posted 2014-01-23 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2018-02

CONDITIONS: Preterm
Keywords: preterm and term newborns; diagnosis of cerebral white matter damage; quantitative brain elasticity; Transfontanel ultrafast doppler
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnosis of white matter damage (Experimental): Added value of supersonic shear imaging in the diagnosis of white matter damage in preterm infants
  Interventions: Other: diagnosis of white matter damage in preterm infants

INTERVENTIONS:
Other: diagnosis of white matter damage in preterm infants — Added value of supersonic shear imaging in the diagnosis of white matter damage in preterm infants

SUMMARY:
Preterm birth and perinatal events related can interrupt microscopic maturation of the developing white matter leading to diffuse injury and subsequent neurocognitive impairments. Brain maturation can be studied using diffusion tensor imaging but is difficult to assess early after birth, repeatedly and at the bedside. Supersonic Shear wave Imaging (SSI) could be of interest in this clinical setting. This technique, already investigated in adults (breast, thyroid or liver fibrosis staging), has not been yet evaluated in neonates.

Objective:

To describe the feasibility and reproducibility of quantitative elasticity mapping in preterm infants and to correlate to gestational age.

Methods:

SSI is a quantitative stiffness imaging technique based on the combination of a remote palpation induced into tissues by the radiation force a focused ultrasonic beam and an ultrafast ultrasound imaging sequence. Such ultrafast frame rates permit to track in real time the displacements induced by the propagation of the resulting shear waves. For each pixel, the shear wave speed can be estimated locally and enables quantitative mapping of the local shear elasticity (characterizing the stiffness in kPa). In this study, we will use a new generation of ultrafast ultrasound scanners (Aixplorer®, Supersonic Imagine, Aix en Provence, France) with a linear L10-2 probe (256 elements, 6 MHz) in neonates born between 25 and 40 weeks' gestation (n=100). Three separate acquisitions will be obtained for each area of interest both on right and left sides and stiffness was measured using a unique ROI of 2.5 cm².

DETAILED DESCRIPTION:
White matter damage occurs in 20% of preterm infants in industrialized countries. These lesions are difficult to evaluate by standard ultrasound. The quantitative elastography is a new medical imaging technique and potentially a diagnostic tool in brain lesions in preterm infants. Shear wave Imaging (SSI) could be of interest in this clinical setting. This technique, already investigated in adults (breast, thyroid or liver fibrosis staging), has not been yet evaluated in neonates.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 24 +0 and 31 +6 j GA) and 39 +0 and 40 +6 d (control group)
* Inborn or Outborn
* Informed consent of the holders of the exercise of parental authority
* recipient of a social security system (excluding AME) Child

Exclusion Criteria:

* Malformation known pathology;
* Known chromosomal abnormality;

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2013-12; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Sequences quantitative elastography and ultra-sensitive Doppler ultrasound performed on AixplorerTM (V2) data of brain MRI preterm infants. | Up to on 40GA + /-1week fo preterm infants<32GA. For newborns at term:on day3+-1d
  To describe the feasibility and reproducibility of quantitative elasticity mapping in preterm infants and to correlate to gestational age
  * For preterm infants <32GA: Quantitative elasticity mapping will be repeated at different stages of postnatal development of preterm infants: on day0-day1, day3 + /-1d, day8, day21 + /-1d; 40GA + /-1week.
  * For newborns at term (39-40GA +6 d) : Quantitative elasticity mapping will be performed on day3+-1

SECONDARY OUTCOMES:
Correlation and comparison of measures elastography MRI to determine the prognosis of brain abnormalities detected by elastography | For preterm infants <32GA:up to 40GA+/-1 week.For newborns at term :on day3+-1
  Longitudinal comparison of measures of quantitative elastography in the supratentorial white matter, corpus callosum, gray matter (basal ganglia) and white matter infratentorial (cerebellar hemispheres) during development in preterm infants <32 weeks and compared the values obtained in the newborn term.
  For preterm infants <32GA:on day0-day1, day3 + /-1d, day8, day21 + /-1d; 40GA + /-1week.For newborns at term :on day3+-1
Quantitative cerebral perfusion values obtained by Doppler ultra-sensitive | up to 40GA + /-1week for preterm infants <32GA .For newborns at term :on day3+-1
  Quantitative cerebral perfusion values obtained by Doppler ultra-sensitive (with standard setting speeds) in premature infants with and without white matter lesions in the frontal white matter and basal ganglia (temporal curve of blood flow in the region interest with defined and standardized measurement of peak systolic and diastolic values: pulsatility index.
Cerebral perfusion values obtained by Doppler ultra-sensitive | on day21 + /-1d
  Cerebral perfusion values obtained by ultra-sensitive Doppler in premature infants with abnormal EEG characterized (positive rolandic spikes> 2 min, convulsions ...) during the first 21 days of life.

CONTACTS AND LOCATIONS:
Overall Officials: Biran Valerie, MP,PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Derived] Faure F, Alison M, Francavilla M, Boizeau P, Guilmin Crepon S, Lim C, Planchette G, Prigent M, Frerot A, Tanter M, Demene C, Baud O, Biran V. Transfontanellar shear wave elastography of the neonatal brain for quantitative evaluation of white matter damage. Sci Rep. 2024 May 23;14(1):11827. doi: 10.1038/s41598-024-60968-w. PMID 38782968